CLINICAL TRIAL: NCT04950283
Title: MR-basierte Charakterisierung Des Knochenmarks in Seiner Bedeutung für Skeletterkrankungen Von Patienten Mit Diabetes
Brief Title: MR-based Characterization of Bone Marrow in Its Relevance to Skeletal Disease in Patients With Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Knoma
Record Dates: First submitted 2021-06-23; First posted 2021-07-06 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2; Osteoporosis; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoporosis; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Magnetic resonance examination and anthropometric, metabolic characterization
  Interventions: Diagnostic Test: magnetic resonance examination, anthropometric and metabolic characterization

INTERVENTIONS:
Diagnostic Test: magnetic resonance examination, anthropometric and metabolic characterization — Participants undergo a magnetic resonance examination, anthropometric characterization and metabolic characterization via oral glucose tolerance test.

SUMMARY:
For a long time, no direct connection was seen between the two common diseases diabetes mellitus and osteoporosis. However, as more and more younger people are affected by obesity, develop type 2 diabetes mellitus and suffer osteoporotic fractures, the question of a connection between these clinical pictures has now arisen.

Modern magnetic resonance imaging and spectroscopy techniques allow detailed and non-invasive characterization of bone marrow in different body regions.

Low body weight (BMI<20kg/m²) has been shown to be associated with decreased bone density, while obesity has long been associated with high cortical bone mass - the idea of bone health. It has now been proven that obesity also has a negative effect on bone structure. Here, it is not only BMI that is crucial, but also the localization of fat tissue in the body. Visceral fat has a directly damaging effect on bone microarchitecture through dysregulated production and release of cytokines and adipokines. Thus, it has been shown that both type 1 and type 2 diabetic patients have a decreased rate of bone remodeling and very obese patients with type 2 diabetes have an increased risk of fracture. It must be concluded that body weight, or BMI, cannot be the sole measure for estimating bone health. Thus, type 2 diabetes shows reduced bone remodeling with normal or slightly increased bone density, but inferior stability. This means that type 2 diabetes is associated with an increased risk of osteoporotic fracture, even when bone density measurements are unremarkable. Loss of trabecular bone structure in red (hematopoietic) bone marrow is also characterized by increasing infiltration of the bone marrow space with fat cells (bone marrow adipose tissue). In contrast, the yellow bone marrow, which is mainly present in the diaphysis of tabular bones, has particularly large amounts of fat incorporated into the reticulum cells.

For a long time, only the role of "placeholder" was attributed to these fat cells, but it has been shown that they interact with other cells via the production of autocrine, paracrine and endocrine hormones and cytokines, or adipokines, and are thus related to the metabolic state of the entire body. A basic assumption here is that the amount of unsaturated fatty acids in the adipose bone marrow is an important and functional marker for different types of adipocytes. It has been shown that 3 individuals with poorer insulin sensitivity have more unsaturated fatty acids in yellow bone marrow.

Thus, the concept of different types of adipocytes in the bone marrow, with their inherent different fatty acid composition could serve to reconcile the at first glance counterintuitive physiological regulation of bone marrow fat and its response to metabolic perturbations.

In order to show whether and how the composition of the yellow (unsaturated fatty acids) and red (bone marrow adipose tissue) bone marrow differs in healthy individuals, individuals with impaired insulin sensitivity in different age groups and patients with type 2 diabetes, and whether this can be used to detect early changes in the bone matrix with regard to bone density, the proportion of bone marrow adipose tissue in the red bone marrow at different locations in the skeleton will be quantified by means of chemical-shift-selective MRI sequences as well as the composition of bone marrow fat in the yellow bone marrow with regard to the proportions of monounsaturated and polyunsaturated fatty acids by means of volume-selective MRS.

A total of 96 healthy volunteers (48 each male and female) aged 25 to 75 years and with body mass index between 18.5 and 35 kg/m² will be included. In addition, 24 patients (12female/12male) with type 2 diabetes will be recruited.

After magnetic resonance examination, anthropometric and metabolic characterization (oral glucose tolerance test) will take place.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18,5 and 35 kg/m²
* Age between 25 and 75 years
* Ability to understand and follow study-related instructions
* Consent to information in case of unexpected detected pathological findings

Exclusion Criteria:

* contraindications for magnetic resonance imaging (metal in or on the body, e.g. pacemaker)
* pregnancy
* people with limited thermal sensors or increased sensitivity to heating
* Persons in whom circulatory disease cannot be excluded after questioning
* Individuals who report a hearing disorder or increased sensitivity to loud sounds
* Claustrophobia
* subjects incapable of giving consent are excluded
* acute illness or infection within the last 4 weeks
* Conditions that, in the judgment of an investigator, jeopardize the success of the study or indicate that the subject is at risk of harm
* type 1 diabetes
* Patients with type 2 diabetes and pharmacologic therapy for diabetes outside of metformin and DPP-IV inhibitors
* HbA1c > 10,0 %
* duration of diabetes >= 2 years

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
monounsaturated and polyunsaturated fatty acids in the yellow bone marrow | about 10 minutes
  The composition of the lipids in the yellow bone marrow (monounsaturated and polyunsaturated fatty acids) will be determined by volume selective Proton magnetic resonance spectroscopy
Fat content in the red bone marrow of the vertebral bodies and femura | 120 seconds
  Proton density fat fraction will be determined by multi-echo Dixon-Imaging
Fat and water selective tomograms from shoulders to knees | 68 seconds
  Fat and water selective tomograms from shoulders to knees will be created by chemical-shift-selective recording technique
Insulin sensitivity | Sample collection will be from 0 to 120 minutes (every 30 minutes)
  Insulin sensitivity will be examined by oral glucose tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Tübingen, Germany